CLINICAL TRIAL: NCT03483675
Title: Randomized Feasibility Study of Discontinuation Versus Continuation of Immunosuppressive Therapy (IST) in Patients With Chronic Graft Versus Host Disease (GVHD)
Brief Title: Discontinuation or Continuation of Immunosuppressive Therapy in Participants With Chronic Graft Versus Host Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Stephanie Lee, Professor and Associate Director, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9962; NCI-2018-00323 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9962 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG1001667 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2018-03-13; First posted 2018-03-30 (Actual); Results first posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Chronic Graft Versus Host Disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Immunosuppression Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (discontinued IST) (Active Comparator): Participants have their IST tapered and discontinued per the plan.
  Interventions: Biological: Immunosuppressive Therapy; Other: Survey Administration
- Arm II (continued IST) (Experimental): Participants continue to receive a fixed dose IST for an additional 9 months with no taper.
  Interventions: Biological: Immunosuppressive Therapy; Other: Survey Administration

INTERVENTIONS:
Biological: Immunosuppressive Therapy — Discontinued IST
  Other Names: Anti-Rejection Therapy; immunosuppression
  Arms: Arm I (discontinued IST)
Biological: Immunosuppressive Therapy — Continued IST
  Other Names: Anti-Rejection Therapy; immunosuppression
  Arms: Arm II (continued IST)
Other: Survey Administration — Ancillary studies

SUMMARY:
This randomized trial studies how well discontinuation or continuation of immunosuppressive therapy works in treating participants with chronic graft versus host disease. Continuation of immunosuppressive treatment may prevent graft-versus-host disease worsening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess feasibility of enrolling and randomizing patients with chronic graft versus host disease (GVHD) to discontinuation (standard of care) versus continuation (investigation) of immunosuppressive therapy (IST).

SECONDARY OBJECTIVES:

I. Assess feasibility of enrolling and randomizing patients who are not local, and evaluate the quality of data received for those patients.

II. Assess whether prolonged IST decreases the need for pulses of high dose IST.

III. Evaluate the effect of prolonged IST on chronic GVHD manifestations and severity, risk of relapse, infection and organ toxicity.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants have their IST tapered and discontinued per the plan.

ARM II: Participants continue to receive a fixed dose IST for an additional 9 months with no taper.

After completion of study treatment, participants are followed up annually.

ELIGIBILITY:
Inclusion Criteria:

* Prior first allogeneic stem cell transplant, with any graft source, donor type, and GVHD prophylaxis
* Patients who are on one systemic immunosuppressive agent for chronic GVHD with a plan to withdraw all systemic IST; hydrocortisone or prednisone continued for treatment of adrenal insufficiency is not considered a systemic IST
* No evidence of malignancy at the time of enrollment
* Agree to be evaluated at the transplant center or by local provider every 3 months for 12 months after randomization
* Agreement to be contacted by phone or e-mail for health status evaluation for up to 3 years
* Signed, informed consent

Exclusion Criteria:

* Inability to comply with study procedures
* Pregancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2021-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Lee, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 participants were not randomized. 1 could not be reached and 3 had a GVHD flare after enrollment.
Period: Overall Study
Arm/Group | Arm I (Discontinued IST) | Arm II (Continued IST)
Started | 9 | 8
Completed | 9 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Discontinued IST) | Arm II (Continued IST) | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 5 | 4 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 9 | 8 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 8 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 8 | 5 | 13
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Enrolling Patients
Description: Descriptive summary of number of patients enrolled on the study (signed consent)
Time Frame: 22.9 months
Measure: Count of Participants; unit: Participants
Groups:
- Total Number of Participants: Total number of participants who signed consent
Arm/Group | Total Number of Participants
Number analyzed (Participants) | 21
Participants | 21

2. Secondary Outcome: Feasibility of Randomizing Patients
Description: Descriptive summary of percentage of patients randomized.
Time Frame: 22.9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Total Number of Participants
Number analyzed (Participants) | 21
Participants | 17

3. Secondary Outcome: Compliance With Treatment
Description: Rate of patients following study immunosuppressive therapy management based on study arm (standard taper or continuation of low dose).
Time Frame: Up to 12 months after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Discontinued IST) | Arm II (Continued IST)
Number analyzed (Participants) | 9 | 8
Participants | 7 | 8

4. Secondary Outcome: Compliance With Data Collection
Description: Count of surveys completed by physicians and patients
Time Frame: Up to 12 months after randomization
Measure: Number; unit: surveys
Arm/Group | Arm I (Discontinued IST) | Arm II (Continued IST)
Number analyzed (Participants) | 9 | 8
surveys
  Total surveys collected | 48 | 39
  Patient surveys missed | 3 | 4
  Physician surveys missed | 5 | 6

5. Secondary Outcome: Graft Versus Host Disease Manifestations
Description: New chronic graft versus host disease (GVHD) manifestations and/or worsening of existing manifestations
Time Frame: Up to 12 months after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Discontinued IST) | Arm II (Continued IST)
Number analyzed (Participants) | 9 | 8
Participants | 2 | 0

6. Secondary Outcome: Recurrent Malignancy
Description: Incidence of relapse of primary disease
Time Frame: Up to 12 months after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Discontinued IST) | Arm II (Continued IST)
Number analyzed (Participants) | 9 | 8
Participants | 0 | 0

7. Secondary Outcome: Incidence of Grade >= 3 Infections
Description: Incidence of grade >= 3 infections
Time Frame: Up to 12 months after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Discontinued IST) | Arm II (Continued IST)
Number analyzed (Participants) | 9 | 8
Participants | 1 | 0

8. Secondary Outcome: Incidence of Grade >= 3 Organ Toxicity
Description: Incidence of grade >= 3 organ toxicity
Time Frame: Up to 12 months after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Discontinued IST) | Arm II (Continued IST)
Number analyzed (Participants) | 9 | 8
Participants | 0 | 0

9. Secondary Outcome: Enrollment Rate of Participants Who Are Not Local
Description: Enrollment rate of participants who are not local. Participants who are local defined as those who had all or some study visits completed at the cancer center.
Time Frame: Up to 12 months after randomization
Population: All participants were local, no data were collected for this outcome measure.
Arm/Group | Arm I (Discontinued IST) | Arm II (Continued IST)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Quality of Data of Participants Who Are Not Local
Description: Participants who are local defined as those who had all or some study visits completed at the cancer center.
Time Frame: Up to 12 months after randomization
Population: All participants were local, no data were collected for this outcome measure.
Arm/Group | Arm I (Discontinued IST) | Arm II (Continued IST)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Arm I (Discontinued IST) | Arm II (Continued IST)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 2/8
Other Adverse Events (participants affected / at risk) | 8/9 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Discontinued IST) (N=9) | Arm II (Continued IST) (N=8)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
heart failure (Cardiac disorders) | 0 (0) | 1 (1) — EF 30%
myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
peripheral ischemia (Vascular disorders) | 0 (0) | 1 (1)
retinal detachment (Eye disorders) | 0 (0) | 1 (1)
stent placement (Cardiac disorders) | 0 (0) | 1 (1)
wound complications (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Arm I (Discontinued IST) (N=9) | Arm II (Continued IST) (N=8)
acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
anal fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
corneal ulcer (Eye disorders) | 1 (1) | 0 (0)
depression (Psychiatric disorders) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
dizziness (General disorders) | 1 (1) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
elevated creatinine (Renal and urinary disorders) | 1 (2) | 0 (0)
essential tremor (Nervous system disorders) | 0 (0) | 1 (1)
fall (General disorders) | 2 (2) | 0 (0)
fatigue (General disorders) | 2/2 (2) | 2 (2)
fecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
fever (General disorders) | 0 (0) | 1 (1)
flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
floaters, eye (Eye disorders) | 0 (0) | 1 (1)
fracture, clavicle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI upset, drug induced (Gastrointestinal disorders) | 0 (0) | 1 (2)
headache (General disorders) | 1 (1) | 0 (0)
hernia, umbilical (Gastrointestinal disorders) | 1 (1) | 0 (0)
hypertriglyceridemia (Gastrointestinal disorders) | 1 (2) | 0 (0)
insomnia (General disorders) | 0 (0) | 2 (2)
iron deficiency anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
IV contrast reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
leukopenia (Immune system disorders) | 2 (2) | 0 (0)
lightheadedness (General disorders) | 1 (1) | 1 (1)
Mucous cyst (toe) (Infections and infestations) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 3 (4) | 1 (1)
neuropathy (Nervous system disorders) | 1 (1) | 2 (2)
prostatitis, presumed (Endocrine disorders) | 1 (1) | 0 (0)
skin, ulcer or lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
skin, erythematous bumps, macules (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
skin, dermatitis, pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
stiffness, muscular (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
urination, difficult (Renal and urinary disorders) | 0 (0) | 1 (1)
weight gain or loss (General disorders) | 1 (1) | 2 (2)
constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
lower respiratory infection (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
phimosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
seizure (Nervous system disorders) | 1 (1) | 0 (0)
thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
thrush (Infections and infestations) | 0 (0) | 1 (1)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 4 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/75/NCT03483675/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/75/NCT03483675/ICF_001.pdf